CLINICAL TRIAL: NCT06150066
Title: Evaluation of the Role of Smoking in the Peri-implantitis Pathogenesis
Brief Title: The Effect of Smoking on Peri-implantitis
Status: Active, not recruiting | Type: Observational
Sponsor: Mustafa Kemal University (Other)
Collaborators: University of Bern (Other); Dokuz Eylul University (Other); Gazi University (Other)
Responsible Party: Principal Investigator, Aysegul SARI, PhD, Assistant professor, Mustafa Kemal University
Other Study IDs: 2023/GOA-8246
Record Dates: First submitted 2023-10-17; First posted 2023-11-29 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Periimplantitis; Microbial Colonization; Cytokines
MeSH Terms: conditions — Peri-Implantitis; Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Smokers with peri-implantitis: 24 patients with smokers with peri-implantitis were included in this group.
  Interventions: Other: Recruiting samples
- Non-smoker individuals with peri-implantitis: 24 patients with non-smokers with peri-implantitis were included in this group.
  Interventions: Other: Recruiting samples
- Smokers with healthy peri-implant tissues: 24 patients with smokers with healthy peri-implant tissues were included in this group.
  Interventions: Other: Recruiting samples
- Non-smoker individuals with healthy peri-implant tissues: 24 patients with non-smokers with healthy peri-implant tissues were included in this group.
  Interventions: Other: Recruiting samples

INTERVENTIONS:
Other: Recruiting samples — The GCF, plaque, and saliva samples will recruited from participants.

SUMMARY:
the primary aim of this project is to evaluate the microbiological and inflammatory effect of smoking status and smoking severity on periimplantitis lesions. The secondary aim is to compare the effect of smoking on periimplantitis and periodontal microbiota and inflammation in the same individuals.

There will include 96 patients, equally divided into four groups: Smokers with peri-implantitis (n=24), non-smoker individuals with peri-implantitis (n=24), smokers with healthy peri-implant tissues (n=24), non-smoker individuals with healthy peri-implant tissues (n=24).

Microbiological and biochemical analyses will be performed on the samples taken.

DETAILED DESCRIPTION:
The cross-sectional study will be carried out in collaboration with the Departments of Periodontology in the Faculty of Dentistry at Bern University, Switzerland, Hatay Mustafa Kemal University, Dokuz Eylul University, Gazi University, and Ege University, Turkey. The first step of the study will be carried out in Turkey, and the second step in Switzerland. Since Hatay is one of the three provinces most affected by the 2023 earthquake in Turkey and Hatay Mustafa Kemal University Dental School was severely damaged, it is impossible to recruit samples from the patients in Hatay. Therefore, this project has been planned as a multicenter, and patient samples will be recruited from the Dokuz Eylül, Gazi University, and Ege University, Department of Periodontology, Faculty of Dentistry. The samples will be analyzed in the Laboratory of Oral Microbiology, Department of Periodontology, University of Bern, Switzerland. The study protocol was approved by the Ethics Committee for the Use of Human Subjects in Research of Dokuz Eylul University (Protocol No: 2023/GOA-8246).

This study will include 96 patients, equally divided into four groups:

* Smokers with peri-implantitis
* Non-smoker individuals with peri-implantitis
* Smokers with healthy peri-implant tissues
* Non-smoker individuals with healthy peri-implant tissues

Smoking status will be categorized into two groups: smoker and non-smoker (never smoker). The non-smoker group will include former smokers who stopped smoking at least 6 years ago.

The cigarettes smoked per day, smoking index (self-reported average cigarettes per day x years of tobacco use), and smoking pocket year will be calculated (self-reported average cigarettes per day x years of tobacco use / the number of cigarettes in a pocket). Smoking status will be detected according to self-report. Smoking status will be later validated by saliva cotinine levels. Salivary cotinine concentration for smoking will be accepted at 5-7 ng/ml. Smoking severity will be determined by higher concentrations.

Periodontal Parameters Clinical periodontal measurements will be assessed using the following for periodontal diagnosis. The measurements will performed using a Williams periodontal probe (Hu-Friedy, Chicago, IL, USA) and include probing pocket depth (PPD), clinical attachment level (CAL), plaque index (PI) 26, gingival index (GI) 27, and percentage bleeding on probing (BOP) 28 at six sites per tooth (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual) on each tooth.

Diagnosis of periodontal diseases and conditions will be made according to the radiographic and clinical diagnostic criteria proposed by the 2017 World Workshop on Classification of Periodontal and Peri-implant Diseases and Conditions.29 Peri-implant health will be assessed by the absence of visual signs of inflammation, bleeding on probing, and further bone loss following initial healing, which should not be ≥2 mm. The criteria for patients with periimplantitis will be PPD≥6 mm in conjunction with profuse bleeding and ≥3 mm bone loss.

Patient demographics and clinical periodontal/peri-implant examination

The following variables will be collected:

* Gender
* Age
* BMI
* Implant age
* Number and location of implants
* Surgical phase steps
* Complications related to implant treatment
* Implant malposition
* Implant Mobility and Discomfort (differences in Periotest values-PTVs)
* Time from loading of implants to current examination (time in function)
* Restorative design
* Prosthesis retention
* Radiographic bone level
* Kind and size of bone defect
* Presence of keratinized mucosa
* Frequency of dental brushing
* Interproximal flossing/brushing
* Frequency of dental appointment
* History of periodontitis
* Reason for tooth loss
* Use of alcohol

Collection of Saliva

Saliva samples will be obtained from patients as unstimulated. Samples will be obtained over 10 min when the participants will be seated. The samples will be kept at -80°C until being transferred to the Department of Periodontology, School of Dental Medicine, University of Bern, in dry ice for the analyses.

Collection of Plaque Samples

Plaque samples will be taken from the periimplantitis and periodontitis subgingival area in the periimplantitis group, and the periodontal healthy and peri-implant health subgingival area in the peri-implant health groups. Subgingival implant and dental plaque samples will be collected from the two deepest periodontal pockets and peri-implant pockets within 200 μl RNAlater in Eppendorf tubes. The sampling sites will be isolated from saliva and slightly air dried. The sample will be collected using a sterile Gracey curette (HuFriedy, Rotterdam, Netherlands). The samples will be taken from the peri-implant health area by the same method in the periimplant health group. Eppendorf microcentrifuge tubes will be stored at -80 °C until being transferred to the Institute of Dentistry, Bern University, in dry ice for the analyses.

Collection of Gingival Crevicular Fluid (GCF) and Peri-implant Sulcus Fluid (PISF) Samples

The samples will be taken from two deepest peri-implant pockets and two deepest periodontal pockets from peri-implantitis patients. Saliva contamination will be avoided by isolating each area with cotton rolls and dehydrating slightly with air. Plaque will be gently removed using a periodontal curette. Using the orifice method, 39 the samples will be obtained within 30 seconds with standardized paper strips (Periopaper; Oraflow Inc., Plainview, NY). The volumes will be measured on a precalibrated electronic gingival fluid measuring device (Oraflow Inc., Plainview, NY). 40 The readings from the electronic device will be converted to an actual volume (μl) by reference to a standard curve. Samples contaminated with blood or saliva will be excluded. All six Periopaper strips will be pooled in plastic Eppendorf microcentrifuge tubes and stored at -80 °C until being transferred to the Institute of Dentistry, Bern University, in dry ice for the analyses.

Laboratory Analyses

Saliva and plaque samples will be transferred to the Laboratory of Oral Microbiology, Department of Periodontology, School of Dental Medicine, University of Bern and all laboratory analyses will be performed by Dr. Aysegul Sari at the Laboratory of Oral Microbiology, Department of Periodontology, School of Dental Medicine, University of Bern, Switzerland after the material transfer agreement is signed.

Biochemical Analysis

Patients' smoking status will be determined by cotinine analysis using an enzyme immunoassay kit in the saliva samples.

Microbiological analysis

The presence and abundance of Fusobacterium nucleatum, Campylobacter rectus, Prevotella intermedia, Aggregatinacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola, Saccharibacteria (TM7), Streptococcus aureus, and Actinomyces oris, will be analyzed in plaque samples. The targeted identification of these bacteria will be made by Real Time Q-PCR. 16sRNA sequencing will be used for an unbiased and untargeted microbiological analysis. Total genomic DNA will be extracted, and then amplification of the 16S rRNA will be performed.

GCF analysis

GCF analysis is planned as a second study. Luminex bead-based multiplex immunoassay will be used to carry out the analysis of GCF and saliva samples. GCF and saliva markers were broadly selected according to previous literature as oxidative stress markers 8-OHdG, PARK7/DJ-1, and NADPH oxidase inflammatory markers IL-1beta, IL-17A/E, osteoprotegerin (OPG); connective tissue degradation markers MMP-8, MMP-3; repair/regeneration markers bone morphogenic protein (BMP)-2, epidermal growth factor (EGF), and vascular endothelial growth factor (VEGF).

Statistical Analysis

Since there is no similar study in the literature, the sample calculation was made on the effect size. The necessary sample size was 24 for each group to detect a significant difference at an effect size (large effect size) of 0.4 and a power level of 90% with a 95% confidence level between the four groups. Gpower package version 3.1 was used for sample size calculations. The normality of continuous variables will be evaluated by Shapiro-Wilk's test. Nonparametric statistical methods will be performed for values with skewed distribution. Kruskal-Wallis test will be performed to compare more than two non-normally distributed variables, and Dunn multiple comparison test for post hoc pairwise multiple comparison analyses. A oneway ANOVA test will be performed to compare more than two normally distributed groups, and the Tukey test will be performed for post hoc pairwise multiple comparison analyses. General linear models will be performed to determine the effect of smoking severity on periimplant and periodontal disease.

ELIGIBILITY:
The inclusion criteria for study groups:

* 18 years old
* Body mass index (BMI) £30 kg/m
* Presence of min 1 implant and 1 tooth for the implant groups
* At least 1 year of implant loading for implant groups for the implant groups

Exclusion criteria for study groups:

* Systemic diseases such as diabetes mellitus, hepatic or renal disease, or other medical conditions or transmittable diseases (ASA score III, IV, V)
* Pregnancy
* Having undergone antibiotics in the previous 6 months
* Periodontal treatment in the previous 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients, who come to the Dokuz Eylül, Gazi, and Ege University, Faculty of Dentistry, Department of Periodontology for routine periodontal control or treatment, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
The evaluation of the abundance of Fusobacterium nucleatum | 2 months
  The presence and abundance of Fusobacterium nucleatum will be analysed by real-time Q-PCR in plaque samples
The evaluation of the abundance of Campylobacter rectus in plaque samples | 2 months
  The presence and abundance of Campylobacter rectus will be analysed by real-time Q-PCR in plaque samples
The evaluation of the abundance of Prevotella intermedia in plaque samples | 2 months
  The presence and abundance of Prevotella intermedia will be analysed by real-time Q-PCR in plaque samplse
The evaluation of the abundance of Aggregatinacter actinomycetemcomitans in plaque samples | 2 months
  The presence and abundance of Aggregatinacter actinomycetemcomitans will be analysed by real-time Q-PCR in plaque samples
The evaluation of the abundance of Porphyromonas gingivalis in plaque samples | 2 months
  The presence and abundance of Porphyromonas gingivalis will be analysed by real-time Q-PCR in plaque samples
The evaluation of the abundance of Tannerella forsythia in plaque samples | 2 months
  The presence and abundance of Tannerella forsythia will be analysed by real-time Q-PCR in plaque samples
The evaluation of the abundance of Treponema denticola in plaque samples | 2 months
  The presence and abundance of Treponema denticola will be analysed by real-time Q-PCR in plaque samples
The evaluation of the abundance of Saccharibacteria (TM7) in plaque samples | 2 months
  The presence and abundance of Saccharibacteria (TM7) will be analyzed by real-time Q-PCR in plaque samplse
The evaluation of the abundance of Streptococcus aureus in plaque samples | 2 months
  The presence and abundance of Streptococcus aureus will be analysed by real-time Q-PCR in plaque samples
The evaluation of the abundance of Actinomyces oris in plaque samples | 2 months
  The presence and abundance of Actinomyces oris will be analysed by real-time Q-PCR in plaque samples

SECONDARY OUTCOMES:
The evaluation of 8-OHdG, PARK7/DJ-1, and NADPH oxidase levels in GCF and saliva samples | 2 months
  The concentrations of 8-OHdG will be analysed by multiplex bead immunoassay method in GCF and saliva
The evaluation of IL-1beta, IL-17A/E, and osteoprotegerin (OPG) levels in GCF and saliva samples | 2 months
  The concentrations of IL-1beta, IL-17A/E, osteoprotegerin (OPG) levels will be analysed by multiplex bead immunoassay method
The evaluation of MMP-8 and MMP-3 levels in GCF and saliva samples | 2 months
  The concentrations of MMP-8, MMP-3 will be analysed by multiplex bead immunoassay method
The evaluation of bone morphogenic protein (BMP)-2, epidermal growth factor (EGF), and vascular endothelial growth factor (VEGF) levels in GCF and saliva samples | 2 months
  The concentrations of bone morphogenic protein (BMP)-2, epidermal growth factor (EGF), and vascular endothelial growth factor (VEGF) will be analysed by multiplex bead immunoassay method

CONTACTS AND LOCATIONS:
Overall Officials: Alpdogan Kantarci, Prof, Study Director — Forsyth Institute; Anton Sculean, Prof, Study Chair — University of Bern; Berrin Unsal, Prof, Study Chair — Gazi University; Aliye Akcali, Prof, Study Chair — Dokuz Eylul University; Aysegul Sari, PhD, Principal Investigator — Mustafa Kemal University
Locations (2):
- University of Bern, Bern, Switzerland
- Hatay Mustafa Kemal University, Antakya, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Derks J, Ichioka Y, Dionigi C, Trullenque-Eriksson A, Berglundh J, Tomasi C, Graziani F. Prevention and management of peri-implant mucositis and peri-implantitis: A systematic review of outcome measures used in clinical studies in the last 10 years. Clin Oral Implants Res. 2023 May;34 Suppl 25:55-67. doi: 10.1111/clr.13925. Epub 2022 Jul 11. PMID 35343614
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] Derks J, Tomasi C. Peri-implant health and disease. A systematic review of current epidemiology. J Clin Periodontol. 2015 Apr;42 Suppl 16:S158-71. doi: 10.1111/jcpe.12334. PMID 25495683
- [Background] Genco RJ. Current View of Risk Factors for Periodontal Diseases. J Periodontol. 1996 Oct;67 Suppl 10S:1041-1049. doi: 10.1902/jop.1996.67.10s.1041. PMID 29539789
- [Background] Roccuzzo A, Stahli A, Monje A, Sculean A, Salvi GE. Peri-Implantitis: A Clinical Update on Prevalence and Surgical Treatment Outcomes. J Clin Med. 2021 Mar 6;10(5):1107. doi: 10.3390/jcm10051107. PMID 33800894
- [Background] Schwarz F, Derks J, Monje A, Wang HL. Peri-implantitis. J Clin Periodontol. 2018 Jun;45 Suppl 20:S246-S266. doi: 10.1111/jcpe.12954. PMID 29926484
- [Background] Curtis MA, Diaz PI, Van Dyke TE. The role of the microbiota in periodontal disease. Periodontol 2000. 2020 Jun;83(1):14-25. doi: 10.1111/prd.12296. PMID 32385883
- [Background] Marsh PD. Microbial ecology of dental plaque and its significance in health and disease. Adv Dent Res. 1994 Jul;8(2):263-71. doi: 10.1177/08959374940080022001. PMID 7865085
- [Background] Buduneli N. Environmental factors and periodontal microbiome. Periodontol 2000. 2021 Feb;85(1):112-125. doi: 10.1111/prd.12355. Epub 2020 Nov 23. PMID 33226700
- [Background] Axelsson P, Paulander J, Lindhe J. Relationship between smoking and dental status in 35-, 50-, 65-, and 75-year-old individuals. J Clin Periodontol. 1998 Apr;25(4):297-305. doi: 10.1111/j.1600-051x.1998.tb02444.x. PMID 9565280
- [Background] de Araujo Nobre M, Mano Azul A, Rocha E, Malo P. Risk factors of peri-implant pathology. Eur J Oral Sci. 2015 Jun;123(3):131-9. doi: 10.1111/eos.12185. Epub 2015 Apr 20. PMID 25894059
- [Background] Koldsland OC, Scheie AA, Aass AM. The association between selected risk indicators and severity of peri-implantitis using mixed model analyses. J Clin Periodontol. 2011 Mar;38(3):285-92. doi: 10.1111/j.1600-051X.2010.01659.x. Epub 2010 Dec 15. PMID 21158898
- [Background] Romandini M, Lima C, Pedrinaci I, Araoz A, Soldini MC, Sanz M. Prevalence and risk/protective indicators of peri-implant diseases: A university-representative cross-sectional study. Clin Oral Implants Res. 2021 Jan;32(1):112-122. doi: 10.1111/clr.13684. Epub 2020 Dec 29. PMID 33210772
- [Background] Farronato D, Azzi L, Giboli L, Maurino V, Tartaglia GM, Farronato M. Impact of Smoking Habit on Peri-Implant Indicators following Different Therapies: A Systematic Review. Bioengineering (Basel). 2022 Oct 18;9(10):569. doi: 10.3390/bioengineering9100569. PMID 36290537
- [Background] Daubert DM, Weinstein BF, Bordin S, Leroux BG, Flemming TF. Prevalence and predictive factors for peri-implant disease and implant failure: a cross-sectional analysis. J Periodontol. 2015 Mar;86(3):337-47. doi: 10.1902/jop.2014.140438. Epub 2014 Nov 21. PMID 25415249
- [Background] Lindquist LW, Carlsson GE, Jemt T. A prospective 15-year follow-up study of mandibular fixed prostheses supported by osseointegrated implants. Clinical results and marginal bone loss. Clin Oral Implants Res. 1996 Dec;7(4):329-36. doi: 10.1034/j.1600-0501.1996.070405.x. PMID 9151599
- [Background] Karoussis IK, Salvi GE, Heitz-Mayfield LJ, Bragger U, Hammerle CH, Lang NP. Long-term implant prognosis in patients with and without a history of chronic periodontitis: a 10-year prospective cohort study of the ITI Dental Implant System. Clin Oral Implants Res. 2003 Jun;14(3):329-39. doi: 10.1034/j.1600-0501.000.00934.x. PMID 12755783
- [Background] Schwarz F, Becker K, Sahm N, Horstkemper T, Rousi K, Becker J. The prevalence of peri-implant diseases for two-piece implants with an internal tube-in-tube connection: a cross-sectional analysis of 512 implants. Clin Oral Implants Res. 2017 Jan;28(1):24-28. doi: 10.1111/clr.12609. Epub 2015 Jul 14. PMID 26178415
- [Background] Bizzarro S, Loos BG, Laine ML, Crielaard W, Zaura E. Subgingival microbiome in smokers and non-smokers in periodontitis: an exploratory study using traditional targeted techniques and a next-generation sequencing. J Clin Periodontol. 2013 May;40(5):483-92. doi: 10.1111/jcpe.12087. Epub 2013 Mar 13. PMID 23489056
- [Background] Zhou N, Huang H, Liu H, Li Q, Yang G, Zhang Y, Ding M, Dong H, Mou Y. Microbiota analysis of peri-implant mucositis in patients with periodontitis history. Clin Oral Investig. 2022 Oct;26(10):6223-6233. doi: 10.1007/s00784-022-04571-1. Epub 2022 Jun 8. PMID 35672515
- [Background] Chih SM, Cheng CD, Chen SH, Sung CE, Huang RY, Cheng WC. The impact of smoking on peri-implant microbiota: A systematic review. J Dent. 2023 Jun;133:104525. doi: 10.1016/j.jdent.2023.104525. Epub 2023 Apr 23. PMID 37088258
- [Background] Tsigarida AA, Dabdoub SM, Nagaraja HN, Kumar PS. The Influence of Smoking on the Peri-Implant Microbiome. J Dent Res. 2015 Sep;94(9):1202-17. doi: 10.1177/0022034515590581. Epub 2015 Jun 29. PMID 26124222
- [Background] Barbagallo G, Santagati M, Guni A, Torrisi P, Spitale A, Stefani S, Ferlito S, Nibali L. Microbiome differences in periodontal, peri-implant, and healthy sites: a cross-sectional pilot study. Clin Oral Investig. 2022 Mar;26(3):2771-2781. doi: 10.1007/s00784-021-04253-4. Epub 2021 Nov 26. PMID 34826030
- [Background] Sari A, Davutoglu V, Bozkurt E, Taner IL, Erciyas K. Effect of periodontal disease on oxidative stress markers in patients with atherosclerosis. Clin Oral Investig. 2022 Feb;26(2):1713-1724. doi: 10.1007/s00784-021-04144-8. Epub 2021 Aug 20. PMID 34415433
- [Background] Yamamoto Y, Nishida N, Tanaka M, Hayashi N, Matsuse R, Nakayama K, Morimoto K, Shizukuishi S. Association between passive and active smoking evaluated by salivary cotinine and periodontitis. J Clin Periodontol. 2005 Oct;32(10):1041-6. doi: 10.1111/j.1600-051X.2005.00819.x. PMID 16174266
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834
- [Background] Caton JG, Armitage G, Berglundh T, Chapple ILC, Jepsen S, Kornman KS, Mealey BL, Papapanou PN, Sanz M, Tonetti MS. A new classification scheme for periodontal and peri-implant diseases and conditions - Introduction and key changes from the 1999 classification. J Periodontol. 2018 Jun;89 Suppl 1:S1-S8. doi: 10.1002/JPER.18-0157. PMID 29926946
- [Background] Araujo MG, Lindhe J. Peri-implant health. J Clin Periodontol. 2018 Jun;45 Suppl 20:S230-S236. doi: 10.1111/jcpe.12952. PMID 29926494
- [Background] Nibali L, Donos N. Periodontitis and redox status: a review. Curr Pharm Des. 2013;19(15):2687-97. doi: 10.2174/1381612811319150003. PMID 23092320
- [Background] Varghese J, Bhat V, Chianeh YR, Kamath V, Al-Haj Husain N, Ozcan M. Salivary 8-hydroxyguanosine levels in smokers and non-smokers with chronic periodontitis. Odontology. 2020 Oct;108(4):569-577. doi: 10.1007/s10266-020-00496-x. Epub 2020 Feb 17. PMID 32065311
- [Background] Sun Q, Shen ZY, Meng QT, Liu HZ, Duan WN, Xia ZY. The role of DJ-1/Nrf2 pathway in the pathogenesis of diabetic nephropathy in rats. Ren Fail. 2016;38(2):294-304. doi: 10.3109/0886022X.2015.1120119. Epub 2015 Dec 7. PMID 26643903
- [Background] Yan YF, Yang WJ, Xu Q, Chen HP, Huang XS, Qiu LY, Liao ZP, Huang QR. DJ-1 upregulates anti-oxidant enzymes and attenuates hypoxia/re-oxygenation-induced oxidative stress by activation of the nuclear factor erythroid 2-like 2 signaling pathway. Mol Med Rep. 2015 Sep;12(3):4734-4742. doi: 10.3892/mmr.2015.3947. Epub 2015 Jun 17. PMID 26081287
- [Background] Di Minno A, Turnu L, Porro B, Squellerio I, Cavalca V, Tremoli E, Di Minno MN. 8-Hydroxy-2-Deoxyguanosine Levels and Cardiovascular Disease: A Systematic Review and Meta-Analysis of the Literature. Antioxid Redox Signal. 2016 Apr 1;24(10):548-55. doi: 10.1089/ars.2015.6508. PMID 26650622